CLINICAL TRIAL: NCT03656575
Title: Reduction of Pro-Inflammatory Synovial Fluid Biomarkers in Osteoarthritis of the Knee With Alpha-2 Macroglobulin: A Randomized Controlled Trial
Brief Title: Reduction of Pro-Inflammatory Synovial Fluid Biomarkers in Osteoarthritis of the Knee With Alpha-2 Macroglobulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-01551
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- intra-articular alpha-2-macroglobulin (Active Comparator): intra-articular injection of 1 mL of the 40 mg/ml strength (1 vial)
  Interventions: Biological: synovial fluid biomarker concentrations
- intra-articular Platelet-rich Plasma (PRP) injection (Active Comparator): Standard of care PRP treatment
  Interventions: Biological: synovial fluid biomarker concentrations
- Intra-articular corticosteroid (Active Comparator): Standard of Care steroid treatment
  Interventions: Biological: synovial fluid biomarker concentrations

INTERVENTIONS:
Biological: synovial fluid biomarker concentrations — Synovial fluid samples will be obtained pre-injection, Post Injection 3 Weeks, Post Injection 6 Weeks, Post Injection 9 Weeks, Post Injection 3 Months, Post Injection 6 Months, Post Injection phone call at 1 Year

SUMMARY:
The purpose of the current study is to assess the ability of alpha-2-macroglobulin treatment to reduce the level of pro-inflammatory synovial fluid biomarkers in patients with osteoarthritis of the knee.

This is a double-blinded rationalized control trial with prospective data collection. The study will collect and analyze the synovial fluid, serum, and urine of patients presenting with knee osteoarthritis in Kellegren-Lawrence grade 2 or 3. It will compare synovial fluid biomarker levels between patients receiving an intra-articular alpha-macroglobulin, intra-articular PR injection and intra-articular corticosteroid serving as a control. Pre-injection pain and function will be assessed. Post-injection pain, function and outcomes will be assessed after six weeks and three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients osteoarthritis classified as Kellegren-Lawrence grade 2 or 3

Exclusion Criteria:

* Mentally impaired (e.g, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Greater than 90 years of age
* Patients with underlying inflammatory arthropathies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Measure of synovial fluid biomarker levels | 6 Weeks
  synovial fluid will be aspirated and analyzed for the presence of 20 biomarkers using bead assay (Milliplex®, Millipore, Billerica MA)
Measure of synovial fluid biomarker levels | 3 Months
  synovial fluid will be aspirated and analyzed for the presence of 20 biomarkers using bead assay (Milliplex®, Millipore, Billerica MA)

CONTACTS AND LOCATIONS:
Overall Officials: Laith Jazrawi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No